CLINICAL TRIAL: NCT04928833
Title: Investigation of the Effects of Pilates Training in Parkinson Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Derya Çağlar, Research Assistant, Recep Tayyip Erdogan University Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2019/10
Record Dates: First submitted 2021-04-27; First posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Parkinson Disease; Pilates; Core Stability; Balance; Quality of Life
Keywords: Parkinson Disease; Pilates; Core Stability; Balance; Quality of Life
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise Movement Techniques; Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Pilates Group (Experimental): Pilates training was carried out as group exercises for about 1 hour, 3 days a week for 8 weeks.
  Interventions: Other: Pilates Training
- Control Group (Active Comparator): Breathing exercises, active range of motion exercises and relaxation exercises were given to the control group as a home program. They were asked to do the exercises 3 days a week for 8 weeks.
  Interventions: Other: Control group
- Evaluation of 'Core' Stability (No Intervention): "Core" stability was evaluated with two important dimensions, "core" strength and endurance tests.
- Ultrasound Examination of M. Transversus Abdominus and M. Multifidus (No Intervention): M. transversus abdominus (TrA) and m. multifidus (MF) muscles were visualized by ultrasonography and the evaluations were performed by an experienced radiologist who was blind to the case groups.
- Evaluation of Lower Extremity Functional Strength (No Intervention): Lower extremity functional strength was evaluated with the 5-Times Sit-and-Stand Test.
- Evaluation of Balance (No Intervention): Balance was evaluated using the Berg Balance Scale (BBS).
- Evaluation of Functional Mobility (No Intervention): Functional mobility was evaluated using the Timed Up and Go Test (TUG).
- Evaluation of Functional Exercise Capacity (No Intervention): Functional exercise capacity was evaluated using the 6 Minute Walking Test (6-MWT).
- Activities of Daily Living and Evaluation of Motor Impairment (No Intervention): Activities of daily living and motor impairment were evaluated with activities of daily living (II) and motor impairment (III) sub-dimensions of the Unified Parkinson's Disease Rating Scale (UPDRS).
- Evaluation of Freezing (No Intervention): The Freezing of Gait Questionnaire (FOGQ) was used to identify and evaluate the subjective perception of Parkinson's patients regarding the severity and effect of freezing on gait performance.
- Evaluation of Fatigue (No Intervention): Fatigue, one of the non-motor findings associated with Parkinson's, was evaluated with the Parkinson's Fatigue Scale-16 (PFS-16).
- Evaluation of Quality of Life (No Intervention): Quality of Life was evaluated with Parkinson's Disease Questionnaire-39 (PDQ-39).

INTERVENTIONS:
Other: Pilates Training — Pilates training was carried out as group exercises for about 1 hour, 3 days a week for 8 weeks. Before starting the exercise training, all subjects were taught the key elements of Pilates in 1 session. Pilates training started with standing exercises for warming up and centering in the supine position. Training continued with upper and lower extremity movements. The intensity of the exercises was increased using different positions and elastic bands. Stretching exercises and posture exercises were used during the cooling period. All exercises were started with 10 repetitions and then increased to 20. In order for the patients to perform the movements correctly, each movement was first demonstrated by the physiotherapist. The movements that the patients could not do were applied by modifying them in a suitable way.
  Arms: Pilates Group
Other: Control group — Breathing exercises, active range of motion exercises and relaxation exercises were given to the control group as a home program. They were asked to do the exercises 3 days a week for 8 weeks.
  Arms: Control Group

SUMMARY:
This study was planned to examine the effects of Pilates training in Parkinson's Patients. The study included 34 Parkinson's patients between Hoehn & Yahr Stage 1-2.5. Pilates training was applied to the Pilates group for 8 weeks, 3 days per week. To the control group; Breathing exercises, active range of motion exercises and relaxation exercises were given as a home program 3 days per week for 8 weeks. It was concluded that Pilates training performed to Parkinson's patients 3 times a week for 8 weeks was effective on "core" stability, thickness of "core" muscles, functional exercise capacity, motor functions, freezing, fatigue and QOL.

DETAILED DESCRIPTION:
This study was planned to examine the effects of Pilates training, which is a "core" stability based exercise method that improves body alignment, postural control and balance, on "core" stability, the thickness of the "core" muscles, functional exercise capacity, motor functions, freezing, fatigue and daily life activities (ADLs) in Parkinson's Patients. The study included 34 Parkinson's patients between Hoehn & Yahr Stage 1-2.5. The patients were randomly divided into two groups as as Pilates (n: 17) and control (n: 17). Pilates training was applied to the Pilates group for 8 weeks, 3 days per week. To the control group; Breathing exercises, active range of motion exercises and relaxation exercises were given as a home program 3 days per week for 8 weeks. The "core" power with the "sit-ups" and the modified "push-ups" tests, the "core" endurans with lateral bridge, trunk flexor endurance and "prone bridge" tests, the thickness of the "core" muscles by ultrasonography, functional strength of the lower limbs with 5 Times Sit Up Test (5TSST), balance with the Berg Balance Scale (BBS), functional mobility; with the Timed Up and Go Test (TUG), functional exercise capacity and walking with the 6-Minute Walk Test (6-MWT), motor impairment with the United Parkinson's Disease Rating Scale (UPDRS)-III, freezing with Freezing of Gait Questionnaire (FOGQ), fatigue with Parkinson's Fatigue Scale (PFS-16), ADLs with UPDRS-II, quality of life (QOL) with Parkinson's Disease Questionnaire-39 (PDQ-39) were evaluated before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* After providing information about the research, agreeing to participate in the research
* Being 40 years or older
* Being diagnosed with '' Idiopathic Parkinson's Disease '' by a specialist
* To be between 1-2.5 values according to Hoehn and Yahr (H&Y) Scale

Exclusion Criteria:

* Standardized Mini Mental Test score is less than 24
* Presence of cardiovascular, pulmonary, orthopedic or other medical conditions that limit participation in Pilates training

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Strength of "Core" Muscles | 8 weeks
  The strength of the trunk muscles was evaluated with 'sit-up' and modified 'push-up' tests. The number of times the subjects could perform each test for 30 seconds was recorded. Each measurement was made twice and the best measurement was used in statistical analysis.
Evaluation of the Endurance of "Core" Muscles | 8 weeks
  Static endurance of the "core" muscles was evaluated using the lateral bridge test defined by McGill, the trunk flexor endurance test and the "prone bridge" test. The time in which the subjects could maintain the test position was recorded in seconds using a stopwatch. Each measurement was made twice and the best measurement was used in statistical analysis. The test was terminated if it disturbed the test position.
Ultrasound Examination of M. Transversus Abdominus and M. Multifidus | 8 weeks
  M. transversus abdominus (TrA) and m. multifidus (MF) muscles were visualized by ultrasonography and the evaluations were performed by an experienced radiologist who was blind to the case groups. Ultrasound recordings were made using B-mode ultrasound. Each measurement was taken 3 times and the average value of 3 measurements was recorded in mm for statistical analysis.
Evaluation of Lower Extremity Functional Strength | 8 weeks
  Lower extremity functional strength was evaluated with the 5-Times Sit-and-Stand Test. The test was performed twice, one trial, and the last measurement was used in statistical analysis.
Evaluation of Balance | 8 weeks
  Balance was evaluated using the Berg Balance Scale (BBS). BBS tests were performed using the materials specified in the directive and in accordance with the instructions. The total score ranges from 0-56, with higher scores indicating better balance.
Evaluation of Functional Mobility | 8 weeks
  Functional mobility was evaluated using the Timed Up and Go Test (TUG). This test; The duration was recorded and applied during the single-task and dual-task (motor and cognitive). Testing for single task was carried out in accordance with the instruction. In dual-motor duty, while holding an empty tray from the case with both hands; In the dual-cognitive task, he was asked to stand up and walk, turn around and come back and sit on the chair, counting 1 each backwards from a certain number (any number from 20 to 100). The time was recorded with a stopwatch. The test was performed twice, one trial, and the last measurement was used in statistical analysis.
Evaluation of Functional Exercise Capacity | 8 weeks
  Functional exercise capacity was evaluated using the 6 Minute Walking Test (6-MWT). The test was performed in accordance with the American Thoracic Society criteria.
  Normal values of 6-MWT are calculated approximately according to age, gender, height and weight in healthy adults. In this study, using reference suggested by Gibbons et al. "Estimated 6-MWT distance" and the rate of reaching the maximal heart rate at the end of 6-MWT were calculated.
Activities of Daily Living and Evaluation of Motor Impairment | 8 weeks
  Activities of daily living and motor impairment were evaluated with activities of daily living (II) and motor impairment (III) sub-dimensions of the Unified Parkinson's Disease Rating Scale (UPDRS). The total score ranges from 0-108, with a higher score indicating a more serious disorder.
Evaluation of Freezing | 8 weeks
  The Freezing of Gait Questionnaire (FOGQ) was used to identify and evaluate the subjective perception of Parkinson's patients regarding the severity and effect of freezing on gait performance. The total score ranges from 0-24, with a higher score meaning that a person's walking performance is more affected by freezing.
Evaluation of Fatigue | 8 weeks
  Fatigue, one of the non-motor findings associated with Parkinson's, was evaluated with the Parkinson's Fatigue Scale-16 (PFS-16). The total score ranged from 16 to 80, and a total of 8 points or more was considered tired.
Evaluation of Quality of Life | 8 weeks
  Quality of Life was evaluated with Parkinson's Disease Questionnaire-39 (PDQ-39). This questionnaire is the most frequently used specific health status measure in PD patients. The total score ranges from 0-100, and lower scores better reflect perceived quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: DERYA CAGLAR, MSc, Study Director — Recep Tayyip Erdogan University Vocational School of Physical Therapy and Rehabilitation
Locations (1):
- Recep Tayyip Erdogan University, Güneysu, Rize Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No